CLINICAL TRIAL: NCT00487474
Title: A Single-Center, Open-Label, Exploratory Study of the Volumizing Effect of Sculptra (Poly-L-lactic Acid) Measured by Three Dimensional Digital Surface Imaging
Brief Title: A Single-Center, Open-Label, Exploratory Study of the Volumizing Effect of SCULPTRA Measured by Three Dimensional Digital Surface Imaging
Status: Completed | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DL6049-0502
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Mid Facial Contour Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sculptra
  Interventions: Device: DL6049 (injectable poly-L-lactic acid)

INTERVENTIONS:
Device: DL6049 (injectable poly-L-lactic acid) — Subjects will be treated with SCULPTRA® every 4-6 weeks in accordance with SCULPTRA® package insert
  Other Names: Sculptra

SUMMARY:
* Measure the mid-facial volumetric correction from SCULPTRA treatment, using three-dimensional digital surface imaging
* Determine the mean change from baseline in facial contour deficiency as measured by the Dermik Nasolabial Photo-numeric Scale
* Correlate volumetric correction with clinical improvement as measured by the Dermik Nasolabial Photo-numeric Scale
* Correlate the mean volumetric change in mid-facial treatment area with the amount of product used
* Evaluate subject and investigator global assessment of improvement and subject treatment satisfaction at the end of treatment
* Obtain photographs pre- and post-treatment for the purpose of providing a subject visual aid during the course of treatment
* Collect safety data

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign a statement of informed consent.
* Subjects must be 18-75 years of age, of any race or gender.
* Female patients of childbearing potential must have a negative urine pregnancy test prior to the first treatment with the product and must use an acceptable form of birth control throughout the study (e.g., oral/systemic contraceptives, an intrauterine device (IUD) or Norplant starting at least 28 days prior to study entry and throughout the study).
* Subjects must display signs of facial contour deficiencies in the area of the nasolabial folds [nasolabial fold scores greater than or equal to 2 (bilaterally) on the Dermik Nasolabial Photo-numeric Scale.
* Subjects must be a suitable candidate for SCULPTRA treatment.
* Subjects must be able to understand the requirements of the study and be willing to comply with the study requirements

Exclusion Criteria:

* Subjects with an allergy to any of the constituents of the product.
* Subjects with a known history of keloids or bleeding disorders.
* Subjects of childbearing potential who are pregnant, or plan to become pregnant within the study timeframe, or who are nursing.
* Subjects with significant facial hair (e.g. mustaches, beards, etc.)
* Subjects with an active inflammatory process or infection in the area to be treated (skin eruptions such as cysts, pimples, rashes, cancerous/pre-cancerous lesions, or any other active skin disease in the treatment area).
* Subjects who plan to undergo major facial surgery [e.g., rhinoplasty (with or without implant), facelift, congenital defect repair, etc.] during the course of the study.
* Subjects who have used or plan to use exclusionary medications/treatments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with signs of facial contour deficiencies in the area of the nasolabial folds [nasolabial fold scores greater than or equal to 2 (bilaterally) on the Dermik Nasolabial Photo-numeric Scale.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Measure the mid-facial volumetric correction from SCULPTRA treatment, using three-dimensional digital surface imaging. | 6 months

SECONDARY OUTCOMES:
Determine the mean change from baseline in Nasolabial volume as measured by 3-D digital surface imaging | 6 months
Correlate volumetric correction with clinical improvement as measured by the Dermik Nasolabial Photo-numeric Scale. | 6 months
Correlate the mean volumetric change in mid-facial treatment area with the amount of product used. | 6 months
Determine mean change from baseline in the contour deficiency score as determined by the investigator. | 6 months
Investigator Global Assessment of Improvement - Excellent Improvement | 6 months
Investigator Global Assessment of Improvement - Much Improved | 6 Months
Investigator Global Assessment of Improvement - Improved | 6 Months
Investigator Global Assessment of Improvement - No Change | 6 Months
Investigator Global Assessment of Improvement - Worse | 6 Months
Subject Global Assessment of Improvement - Excellent Improvement | 6 Months
Subject Global Assessment of Improvement - Much Improved | 6 Months
Subject Global Assessment of Improvement - Improved | 6 Months
Subject Global Assessment of Improvement - No Change | 6 Months
Subject Global Assessment of Improvement - Worse | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, MT, ASCP, Study Director — Sanofi
Locations (1):
- London, United Kingdom